CLINICAL TRIAL: NCT06242938
Title: Early Intensive Antihypertensive Treatment in High-risk Population of Intracerebral Hemorrhage Expansion Predicted by Artificial Intelligence
Acronym: ARCHES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Na Li, Principal Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARCHES
Record Dates: First submitted 2023-12-03; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intensive antihypertensive treatment group (Experimental): 1. Treatment starts within 1 hour after randomization
  2. SBP target:130-140 mmHg within 1 hour after treatment
  3. Under the guidance of medication, the researchers can independently select oral + intravenous antihypertensive medications
  Interventions: Procedure: Early intensive antihypertensive treatment
- Standard antihypertensive treatment group (No Intervention): 1. Empirical antihypertensive treatment
  2. SBP target: 140-180 mmHg after randomization

INTERVENTIONS:
Procedure: Early intensive antihypertensive treatment — 1. Treatment starts within 1 hour after randomization
  2. SBP target:130-140 mmHg within 1 hour after treatment
  3. The researchers can independently select oral + intravenous antihypertensive medications. Any type of antihypertensive drugs can be selected (eg. β-blokers, α-blockers, CCBs, ARBs/ACEIs, diuretic, etc.).
  Arms: Early intensive antihypertensive treatment group

SUMMARY:
The goal of this clinical trial is to clarify the efficacy, safety and feasibility of early intensive antihypertensive treantment in intracerebral hemorrhage (ICH) patients at high risk of hematoma expansion based on artificial intelligence prediction.

The main question it aims to answer are:

* Can ICH patients at high risk of hematoma expansion based on artificial intelligence prediction benefit from early intensive antihypertensive treatment?
* Is early intensive antihypertensive treatment safe to patients at high risk of hematoma expansion based on artificial intelligence prediction.

Participants will accept intensive antihypertensive treatment (target systolic blood pressure: 130-140mmHg) at early stage (within 1 hour after randomization) of cerebral hemorrhage and maitain the target blood pressure for 7 days.

Researchers will compare standard treatment group (target systolic blood pressure 140-180mmHg after randomization) to see if intensive antihypertensive treatment can improve the outcome of patients with ICH.

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥ 18 years;
* ② Arrival at the hospital within 6h of onset, able to complete randomization and receive antihypertensive treatment within 1h of arrival (if the time of onset is unclear, the last normal time will be used);
* ③ CT-confirmed spontaneous supratentorial brain parenchymal hematoma that can break into the ventricles and subarachnoid space, with a hematoma volume of <60 ml;
* ④ Patients at high risk of hematoma expansion with ≥3 points on the artificial intelligence-based hematoma expansion 5-point prediction score;
* ⑤ GCS >8;
* ⑥ SBP in the range of 150-220 mmHg after onset and before randomization;
* ⑦ Signed informed consent by the patient or legal representative.

Exclusion Criteria:

* ① Cerebral hemorrhage is caused by known secondary causes such as trauma, tumors, cerebrovascular malformations, and thrombolysis and thrombus extraction
* ② When the brain parenchyma hemorrhage involves the ventricles, the blood completely fills one lateral ventricle or more than half of both lateral ventricles.
* ③ The hematoma of previous intracerebral hemorrhage has not yet been absorbed
* ④ Surgical treatment is planned within 24 hours
* ⑤ Combination of conditions known to be inappropriate for intensive blood pressure lowering (e.g., severe carotid artery stenosis, vertebral artery or intracranial artery stenosis, smoky or Takayasu's arteritis, and severe heart valve stenosis)
* ⑥Combination of known well-defined indications requiring a more aggressive antihypertensive treatmenr, such as hypertensive encephalopathy or aortic coarctation
* ⑦ Known allergy to antihypertensive drugs
* ⑧Known allergy to antihypertensive drugs (i.e., warfarin with INR > 1.5 or other anticoagulant drugs within the past 24 hours).
* ⑨ With platelet counts less than 50,000/mm3.
* ⑩ Disability due to prior illness mRS ≥ 3
* ⑪ Pregnancy status or within 30 days after delivery
* ⑫ Severe heart or liver disease, severe renal insufficiency (eGFR <30 ml/min) or malignant tumor with life expectancy <3 months.
* ⑬ Currently participating in other interventional clinical trials
* ⑭ Informed consent cannot be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Death or severe disability (modified Rankin Scale 3-6) at 90 days | 90 days
  Death or severe disability is defined as modified Rankin Scale (mRS) 3-6. The mRS is a scale used to measure the degree of disability caused by stroke or other neurological conditions. It ranges from 0 (no symptoms) to 6 (death). The lower the score, the less severe the disability.

SECONDARY OUTCOMES:
Hematoma expansion within 24 hours | 24 hours
  Hematoma volume increase ≥6ml on follow up non-contrast CT.
Early neurological deterioration (END) within 24h | 24 hours
  Within 24 hours after onset, NIHSS increase ≥4 or GCS decreased ≥2 (compared to baseline);
Modified Rankin Scale (mRS) distribution at 90 days | 90 days
  The mRS is a scale used to measure the degree of disability caused by stroke or other neurological conditions. It ranges from 0 (no symptoms) to 6 (death). The lower the score, the less severe the disability.
Death at 90 days | Up to 90 days
EuroQol-5 Dimensions (EQ-5D) score at 90 days | 90 days
  The EQ-5D is a standardized instrument for measuring generic health status developed by the EuroQol Group. It assesses five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels: no problems, some problems, and severe problems. The EQ-5D scores range from -0.594 to 1, where 1 represents full health and 0 represents death. Lower scores indicate poorer health. The EQ-5D is commonly used in economic evaluations of health care interventions to assess quality-adjusted life years (QALYs).
Death or severe disability (modified Rankin Scale 3-6) at 180 days | Up to 180 days
  Death or severe disability is defined as modified Rankin Scale (mRS) 3-6. The mRS is a scale used to measure the degree of disability caused by stroke or other neurological conditions. It ranges from 0 (no symptoms) to 6 (death). The lower the score, the less severe the disability.

OTHER OUTCOMES:
Severe hypoperfusion event | Up to 180 days
  Including acute kidney injury, severe hypotension, oliguria, acute myocardial infarction, acute cerebral infarction, etc.
Treatment-related serious adverse events (SAEs) during hospitalization | During hospitalization
Death during hospitalization | During hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Kaijiang Kang, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No